CLINICAL TRIAL: NCT02049333
Title: Phacoemulsification Versus Phacoemulsification With Endoscopic Cycloplasty (ECPL) for Treatment of Plateau Iris Configuration or Syndrome: A Prospective Randomized Clinical and Surgical Study
Brief Title: Cataract Surgery vs Cataract Surgery With ECPL for Treatment of Plateau Iris Configuration or Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Credit Valley EyeCare (Industry)
Responsible Party: Principal Investigator, Iqbal Ike Ahmed, MD, Credit Valley EyeCare
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ECPLateau10.1
Record Dates: First submitted 2014-01-27; First posted 2014-01-30 (Estimated); Last update posted 2014-01-30 (Estimated); Status verified 2014-01

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Phacoemulsification

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phacoemulsification (Active Comparator): Cataract extraction alone
  Interventions: Procedure: Phacoemulsification
- Phacoemulsification with Endoscopic Cycloplasty (ECPL) (Experimental): Cataract extraction combined with endoscopic cycloplasty
  Interventions: Procedure: Phacoemulsification; Procedure: Endoscopic Cycloplasty (ECPL)

INTERVENTIONS:
Procedure: Phacoemulsification
Procedure: Endoscopic Cycloplasty (ECPL)
  Arms: Phacoemulsification with Endoscopic Cycloplasty (ECPL)

SUMMARY:
The purpose of this study is to assess and compare the mechanical angle opening in patients with angle closure due to a plateau iris configuration (elevated iris) using phacoemulsification combined with endoscopic cycloplasty versus treatment with phacoemulsification alone.

ELIGIBILITY:
Inclusion Criteria:

* Patient has to be ≥ 18 years of age of either gender
* Nuclear sclerotic cataract graded by LOCS III to be < 5
* Diagnosis of Plateau Iris Configuration or Syndrome
* No contraindication for cataract or ECPL operation
* Written informed consent on IRB approved Informed Consent Form

Exclusion Criteria:

* Hard cataracts, LOCS III 5 and 6
* Ciliary body cysts
* Clinically significant sequelae from trauma in which angle anatomy/physiology may have been compromised (e.g., chemical burns, significant angle recession, blunt trauma, etc.)
* Congenital anomaly of the irido-trabecular angle
* Previous intraocular surgery
* Previous laser gonioplasty to either eye
* Placement of the intraocular lens in any place other than the capsular bag
* Pupilloplasty
* Rubeosis
* Peripheral anterior synechiae (PAS) nasal angle and/or >180 degrees of PAS
* Neovascular glaucoma; or glaucoma associated with vascular ischemic disorders
* Active corneal inflammation or edema (e.g., keratitis, keratoconjunctivitis, keratouveitis)
* Corneal opacities or disorders that would inhibit visualization of the nasal angle
* Chronic ocular inflammatory disease or presence of active ocular inflammation with risk for synechial/proliferative changes
* Inability to attend regular follow-up assessment or to give informed written consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-11; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Anterior Chamber Angle Depth (nasal angle) | Twelve months
  Anterior chamber angle depth (nasal angle) measured using the Shaffer grading system and via anterior segment imaging

SECONDARY OUTCOMES:
Number of glaucoma medications | Twelve months post-op
  The number of glaucoma medications will be recorded and compared to pre-operative number of glaucoma medications.
Intraocular pressure (IOP) | Twelve months post-op
  IOP will be recorded and compared to pre-operative IOP.

OTHER OUTCOMES:
Intra- and post-operative complications | Up to one year after surgery
  Analyzing any unexpected complications from the surgery such as prolonged hypotony, intraocular pressure spike, prolonged corneal inflammation etc. This will be done during the clinic visit and analyzed under slit lamp examination.

CONTACTS AND LOCATIONS:
Overall Officials: Ike K Ahmed, MD FRCSC, Study Director — University of Toronto, Toronto, Canada
Locations (2):
- Canada (2):
  - Osler EyeCare, Brampton, Ontario
  - Credit Valley EyeCare, Mississauga, Ontario